CLINICAL TRIAL: NCT06242847
Title: Role of Insulin Action in Psoriasis Pathogenesis
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Other Study IDs: AAAU4674
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis; Plaque Psoriasis; Insulin Resistance; PreDiabetes; Overweight and Obesity
Keywords: Insulin; Insulin resistance; Psoriasis
MeSH Terms: conditions — Psoriasis; Insulin Resistance; Prediabetic State; Overweight; Obesity | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood samples during OGTT: fasting and at 120 min after ingestion of 75 g of glucose
  * Skin punch biopsies of lesional (psoriatic) and non-lesional skin taken while fasting and at 120 min after ingestion of 75 g glucose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Insulin Sensitive (IS) with psoriasis: Patients with plaque psoriasis found to have:
  * Hemoglobin A1c < 5.7%
  * Fasting plasma glucose: < 95 mg/dL
  * Fasting serum insulin: < 10 micro-international units per milliliter (μIU/mL)
  * 2-hour post-challenge glucose < 140 mg/dL
  NOTE: Group assignments made retroactively based on the observational study results.
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Procedure: Skin punch biopsy
- Insulin Intermediate (II) with psoriasis: Patients with plaque psoriasis found to have:
  * Hemoglobin A1c < 6.5%
  * Fasting plasma glucose <125 mg/dL
  * Fasting serum insulin: <15 μIU/mL
  * 2-hour post-challenge glucose < 200 mg/dL
  NOTE: Group assignments made retroactively based on the observational study results.
  • Not otherwise meeting all criteria for inclusion in the IS group
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Procedure: Skin punch biopsy
- Insulin Resistant (IR) with psoriasis: Patients with plaque psoriasis found to have:
  * Fasting serum/plasma insulin ≥ 15 μIU/mL
  * Fasting plasma glucose 80-125 mg/dL and
  * Hemoglobin A1c < 6.5% and
  * 2-hour post-challenge glucose < 200 mg/dL
  NOTE: Group assignments made retroactively based on the observational study results.
  Interventions: Diagnostic Test: Oral glucose tolerance test (OGTT); Procedure: Skin punch biopsy

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test (OGTT) — Participants ingest 75 g of glucose in 10 fl oz aqueous solution (fruit flavored) after an overnight fast. Blood is drawn at baseline (t = 0 min) and at 120 min after ingestion. This test is non-experimental.
Procedure: Skin punch biopsy — Punch biopsies are taken from lesional (psoriatic) and non-lesional skin after an overnight fast and at 120 min after ingestion of glucose during OGTT. This procedure is non-experimental.

SUMMARY:
The goal of this study is to collect more information from people with plaque psoriasis and to determine if insulin plays a role in the pathogenesis of psoriasis. The main question it aims to answer is if insulin action is preserved or even enhanced in psoriatic lesions despite insulin resistance elsewhere. Participants with plaque psoriasis will have punch biopsies taken of lesional and non-lesional skin after an overnight fast and then during an oral glucose tolerance test. Biopsy specimens will then be assessed for markers of insulin action.

DETAILED DESCRIPTION:
Psoriasis exhibits a clear and robust epidemiologic association with type 2 diabetes mellitus (T2DM). Although T2DM may exacerbate psoriasis and/or complicate its treatment, we do not understand the mechanisms connecting them. As a starting point, psoriasis appears to worsen the insulin resistance (IR) that underlies T2DM. The study investigators hypothesize that the hyperinsulinemia that attempts to compensate for IR retains the ability to drive proliferation of psoriatic lesions. This would set up a vicious cycle in which psoriasis worsens IR, which in turn stimulates insulin hypersecretion that further intensifies psoriasis. In order to test this hypothesis, the investigators must first determine if insulin signaling in psoriatic lesions is actually hyperactive. The investigators therefore propose in this pilot study to elucidate the nature of insulin signaling in psoriasis by measuring phosphorylation of AKT, insulin's key intracellular signaling mediator, in skin biopsies. We will perform shave punch biopsies of lesional and non-lesional skin in overnight-fasted patients with psoriasis who are overweight or obese and therefore at risk of IR. Another set of biopsies will be taken during an oral glucose tolerance test that stimulates endogenous insulin secretion. The investigators expect that AKT phosphorylation will be attenuated in non-lesional skin of patients determined to have IR compared to those who are Insulin Sensitive (IS) or Insulin Intermediate (II), but that AKT phosphorylation will be preserved or even enhanced in lesional skin despite IR. Determining that insulin action is excessive in psoriatic lesions would suggest reducing insulin levels as a novel psoriasis treatment strategy that would also help to spare patients from difficult immunomodulatory treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index of 25.0-40.0 kg/m2
2. Able to understand written and spoken English and/or Spanish
3. Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.
4. Diagnosed with plaque psoriasis, documented using Psoriasis Area and Severity Index (PASI)
5. Glucose metabolism status as follows (determined only retrospectively based on data collected during the study):

   * For Insulin Sensitive (IS) group:

     • Hemoglobin A1c < 5.7%, and
     * Fasting plasma glucose < 95 mg/dL, and
     * Fasting plasma insulin < 10 μIU/mL, and
     * 2-hour post-challenge glucose < 140 mg/dL
   * For Insulin Intermediate (II) group:

     • Hemoglobin A1c < 6.5%, and

     • Fasting plasma glucose 80-125 mg/dL, and

     • Fasting plasma insulin < 15 μIU/mL, and

     • 2-hour post-challenge glucose < 200 mg/dL, and

     • Not otherwise meeting all criteria for the IS group
   * For Insulin Resistant (IR) group:

     * Hemoglobin A1c < 6.5%, and
     * Fasting plasma glucose 80-125 mg/dL, and
     * Fasting plasma insulin ≥ 15 μIU/mL, and
     * 2-hour post-challenge glucose < 200 mg/dL

NOTE: Group assignments will be made retroactively, after observational data has been collected. Those not fitting into any of these groups will have their data excluded from further analysis.

Exclusion Criteria:

1. Inability to provide informed consent in English or Spanish
2. Laboratory evidence of diabetes mellitus, either determined during the study or based on previous documentation:

   • Hemoglobin A1c ≥ 6.5%, and/or
   * Fasting plasma glucose ≥ 126 mg/dL
   * Plasma glucose ≥ 200 mg/dL at 2 hours after ingestion of a 75-g oral glucose load
   * Random plasma glucose ≥ 200 mg/dL associated with typical hyperglycemic symptoms, diabetic ketoacidosis, or hyperglycemic-hyperosmolar state
3. History of gestational diabetes mellitus
4. Use of antidiabetic medications within the 90 days prior to screening, including those prescribed for other indications (e.g., weight control, restoration of ovulation in of polycystic ovarian syndrome), including:

   • Metformin, thiazolidinediones, sulfonylureas, meglitinides, dipeptidyl peptidase-4 (DPP4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists, sodium/glucose cotransporter 2 (SGLT2) inhibitors, amylin mimetics, acarbose, insulin
5. Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease)
6. Reproductive concerns

   i. Women of childbearing potential not using highly effective contraception, defined as:

   • Surgical sterilization (e.g., bilateral tubal occlusion, bilateral oophorectomy and/or salpingectomy, hysterectomy)

   • Combined oral contraceptive pills taken daily, including during the study

   • Intrauterine device (levonorgestrel-eluting or copper) active at the time of the study
   * Medroxyprogesterone acetate (Depo-Provera®) injection active at the time of the study
   * Etonogestrel implants (e.g., Implanon®, etc.) active at the time of the study
   * Norelgestromin/ethinyl estradiol transdermal system (e.g., Ortho-Evra®) active at the time of the study NOTE: Women not using any of the above forms of birth control may be included if they have a negative urine pregnancy test on the day of the study, before beginning any study procedures.

   ii. Women currently pregnant

   iii. Women currently breastfeeding
7. Known, documented history, at the time of screening, of any of the following medical conditions:

   i. Bleeding disorders, including due to anticoagulation or use of P2Y12 inhibitors ii. Anemia requiring treatment iii. Glucose-6-phosphate dehydrogenase (G6PD) deficiency
8. Use of medications associated methemoglobinemia within 48 hours of shave biopsy procedures:

   i. Nitrates/nitrites: nitric oxide, nitroglycerin, nitroprusside, nitrous oxide ii. Antineoplastics: cyclophosphamide, flutamide, hydroxyurea, ifosfamide, rasburicase iii. Antibiotics: dapsone, nitrofurantoin, paraaminosalicylic acid, sulfonamides iv. Antimalarials: chloroquine, primaquine v. Anticonvulsants: phenobarbital, phenytoin, valproic acid vi. Others: acetaminophen, metoclopramide, quinine, sulfasalazine
9. History of severe infection or ongoing febrile illness within 30 days of screening
10. Any other disease, condition, or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.

13. Known allergy/hypersensitivity to any component of the medicinal product formulations (including amide anesthetics), IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.

14. Concurrent enrollment in another clinical study of any investigational drug therapy within 6 months prior to screening or within 5 half-lives of an investigational agent, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with plaque psoriasis but without diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Skin insulin sensitivity: ratio of phosphorylated to total AKT in skin biopsies | Up to 120 minutes from the start of OGTT
  Investigators will perform Western blots on skin biopsies using antibodies to phosphorylated (T308, S473) and total AKT. The ratio of phosphorylated to total AKT will be determined using densitometry of Western blots and/or by enzyme-linked immunosorbent assays (ELISA), each measured in arbitrary units (AU).

SECONDARY OUTCOMES:
Serum triglyceride (TG) level during OGTT | During OGTT (up to 120 minutes from start of OGTT)
  Measurement of serum triglyceride level (units: mg/dL) during OGTT. A blood test will be done.
Serum free fatty acid (FFA) levels during OGTT | During OGTT (up to 120 minutes from start of OGTT)
  Measurement of serum free fatty acid levels (units: mmol/L) during OGTT. A blood test will be done.
Fasting plasma glucose level | Before OGTT (baseline = 0 minutes), During OGTT (up to 120 minutes from start of OGTT)
  Plasma glucose (units: mg/dL) after an overnight fast (> 8 hours). A blood test will be done. A healthy (normal) fasting blood glucose level for someone without diabetes is 70 to 99 mg/dL.
Fasting serum insulin level | Before OGTT (baseline = 0 minutes), During OGTT (up to 120 minutes from start of OGTT)
  Serum insulin (units: μIU/mL) after an overnight fast (> 8 hours). A blood test will be done. The normal range of fasting insulin varies somewhat between labs, but around 2 to 20 mIU/mL is considered normal by most.
Fasting serum C-peptide level | Before OGTT (baseline = 0 minutes), During OGTT (up to 120 minutes from start of OGTT)
  Serum C-peptide (units: ng/mL) after an overnight fast (> 8 hours). A blood test will be done. A normal result of a C-peptide test ranges from 0.5 ng/mL to 2.0 ng/mL (or 0.17 to 0.83 nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided